CLINICAL TRIAL: NCT00001102
Title: Metabolic Consequences of Highly Active Antiretroviral Therapy (HAART) in HIV-Positive Individuals
Brief Title: The Effect of Anti-HIV Therapy on Fat Metabolism in HIV-Positive Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CPCRA 061; 11616 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Body Composition; Anti-HIV Agents; Cholesterol; Triglycerides
MeSH Terms: conditions — HIV Infections

SUMMARY:
The purpose of this study is to see how taking certain anti-HIV drugs affects the way the body metabolizes fat. This study will evaluate patients who are enrolled in CPCRA 058 (the FIRST [Flexible Initial Retrovirus Suppressive Therapies] study) by looking for changes in cholesterol levels, levels of fat in the blood, and body fat distribution. Patients in the FIRST study receive an anti-HIV drug regimen which contains a protease inhibitor (PI), a nonnucleoside reverse transcriptase inhibitor (NNRTI), or both.

Anti-HIV drug therapy using PIs has become very common treatment for HIV-positive patients. Recently, however, serious side effects involving how the body uses fat are being reported in patients taking PIs. Examples of these side effects are a redistribution of body fat, high cholesterol level, and development of diabetes. However, some of these side effects have also been seen in patients who are not taking PIs. It is important to determine whether or not these side effects are directly related to PI use. In this study, patients on different drug combinations, either with or without a PI, will be compared.

DETAILED DESCRIPTION:
Close to 3 years into widespread PI use, several toxicities, including metabolic alterations, are being reported increasingly in conjunction with the use of PI-containing regimens. Some of the manifestations of these metabolic alterations include hyper/dyslipidemia, hyperglycemia, insulin resistance and glucose intolerance, lipodystrophy (in face and extremities), and body fat redistribution (e.g., central obesity and buffalo humps). Despite reports of increasing prevalence of metabolic complications among PI users, the question of whether they result from PI therapy has not been answered. Some of these complications, e.g., a decrease in peripheral fat with an increase in visceral fat and buffalo hump, have been observed in HIV-infected individuals who were not receiving PIs. This study compares 3 different antiretroviral regimens used in the FIRST study (CPCRA 058), 1 of which does not contain a PI, and examines metabolic alterations which occur.

This study enrolls patients simultaneously co-enrolling in the FIRST protocol; 120 patients from each of the FIRST study strategy groups. At entry, Months 1 and 4, and then every 4 months, blood is drawn to measure serum glucose, insulin, total cholesterol, HDL cholesterol, LDL cholesterol, and triglyceride levels. At entry and Months 4, 8, 12, and then every 12 months, body cell mass, and body fat by bioelectrical impedance analysis (BIA) are assessed. [AS PER AMENDMENT 7/5/01: At Months 4, 8, and 12, then every 4 months through closure of the FIRST protocol] patients are weighed and skinfold measurements and body circumference measurements are done. The skinfold and body circumference measurements will be discontinued after the study has collected a minimum of 2 years of follow-up data on all participants. Statistical evaluations are performed on the data.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are enrolled in the FIRST study (CPCRA 058).
* Have written informed consent of parent or guardian if under the age of 18.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 460
Dates: Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subha Raghavan, Study Chair
Locations (15):
- United States (15):
  - Community Consortium / UCSF, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Wayne State Univ - WSU/DMC / Univ Hlth Ctr, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners in Research / New Mexico, Albuquerque, New Mexico
  - Harlem AIDS Treatment Grp / Harlem Hosp Ctr, New York, New York
  - The Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium / Div of Infect Diseases, Richmond, Virginia

REFERENCES:
- [Result] Visnegarwala F, Chen L, Raghavan S, Tedaldi E. Prevalence of diabetes mellitus and dyslipidemia among antiretroviral naive patients co-infected with hepatitis C virus (HCV) and HIV-1 compared to patients without co-infection. J Infect. 2005 May;50(4):331-7. doi: 10.1016/j.jinf.2004.06.001. PMID 15845431
- [Result] Visnegarwala F, Shlay JC, Barry V, Gibert CL, Xiang Y, Wang J, Kotler D, Raghavan S, El-Sadr WM; for Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA). Effects of HIV infection on body composition changes among men of different racial/ethnic origins. HIV Clin Trials. 2007 May-Jun;8(3):145-54. doi: 10.1310/hct0803-145. PMID 17621461